CLINICAL TRIAL: NCT02012465
Title: Validation of Insulin Protocol for Prevention and Management of Hyperglycemia in Oncology Patients With Diabetes Receiving High Dose Glucocorticoid Therapy
Brief Title: Validation of Insulin Protocol for Glucocorticoid-induced Hyperglycemia in Diabetic Oncology Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201306071
Record Dates: First submitted 2013-12-02; First posted 2013-12-16 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma; Diabetes Mellitus, Type 2; Hyperglycemia
Keywords: Steroid induced hyperglycemia; Glucocorticoid induced hyperglycemia
MeSH Terms: conditions — Lymphoma; Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin protocol (Experimental): For diabetic patients, as part of the initial chemotherapy orders on admission, the following will be calculated by the primary oncologist to determine the amount of neutral protamine Hagedorn (NPH) insulin needed to cover steroid use in prednisone equivalents (all insulin in this study is to be administered subcutaneously):
  * Use 0.1 (mg of prednisone equivalent - 20)/20 x weight (kg) to estimate total insulin in 24 hours (Total daily dose (TDD))
  * Total daily NPH dose will be divided equally based on the frequency of steroid administration, and given with each steroid dose.
  For nondiabetic participants with hyperglycemia recruited during admission, the inpatient oncology team will consult the endocrine team within 24 hours of eligibility for NPH dosing as above.
  Interventions: Biological: Insulin protocol

INTERVENTIONS:
Biological: Insulin protocol — Within 24 hours of admission for diabetic participants, the inpatient oncology team will consult the endocrine team to apply the following part of the protocol, confirm NPH insulin dosing, and ensure that oral hypoglycemics are held.
  The following basal-bolus protocol is standard of care for inpatient diabetics requiring insulin at Barnes Jewish Hospital. The alternative practice has been to use 60-80% of the home insulin regimen while patients are hospitalized. For patients using home insulin, the admitting oncology team will enact one of these methods while awaiting the endocrine service's formal recommendations.
  * Determine basal-bolus insulin requirement for the patient based on body weight: Patient weight (kg) x 0.5-0.7 Units/kg = Units of total insulin per 24 hours
  * The TDD can be divided into 50% basal (glargine) and 50% meal time (lispro) insulin, plus sliding scale insulin (lispro).
  Other Names: NPH; Glargine; Lispro

SUMMARY:
There are no guidelines for the management of glucocorticoid- (henceforth steroid) induced elevated blood sugars (henceforth hyperglycemia). Oncology ward patients have particularly high rates of hyperglycemia and are frequently exposed to high dose steroid therapy. A prior study by Muthala et al. (unpublished data) found a relationship between insulin requirements needed to maintain normal blood sugars, patient weight, and mg of steroid administered. In this pilot study, through an endocrine consult team, a weight-based, steroid dose-based insulin protocol will be implemented for the management of hyperglycemia in lymphoma patients requiring high dose steroid therapy, with the goal of reducing hyperglycemia incidence.

ELIGIBILITY:
For diabetics enrolled on admission:

Inclusion Criteria:

* Age ≥ 18 years old
* Type 2 diabetes mellitus treated with insulin secretagogues or insulin prior to hospitalization
* Diagnosis of lymphoma
* Plan to treat with steroids of minimum equivalent of 20 mg prednisone per day
* Hospitalized for at least 48 hours
* Decision-making capacity to provide own consent

Exclusion Criteria:

* Type 1 diabetes
* Any contraindication to insulin therapy
* Patients only on single agent therapy such as metformin, thiazolidinediones (TZDs), Dipeptidyl peptidase-4 (DPP4) inhibitors, or Exenatide®, for safety concerns
* Insulin requirement of >1.5 units of insulin/kg
* If a patient required ICU stay during the hospitalization, data from 12 hours before, during, and 12 hours after ICU stay will be omitted to avoid confounding of the effect of critical illness on glycemic control
* Pregnancy, confirmed with a urine b-human chorionic gonadotropin (HCG) (for all women between the age of 18 and 60 years old)

Patients who develop a blood glucose > 235 mg/dL after admission will be eligible for study enrollment based on the following:

Inclusion criteria:

* Age ≥ 18 years old
* Diagnosis of lymphoma
* Plan to treat with steroids of minimum equivalent of 20 mg prednisone per day
* Will be hospitalized for at least an additional 48 hours
* Decision-making capacity to provide own consent

Exclusion criteria:

* Any contraindication to insulin therapy
* If a patient required ICU stay during the hospitalization, data from 12 hours before, during, and 12 hours after ICU stay will be omitted to avoid confounding of the effect of critical illness on glycemic control
* Pregnancy, confirmed with a urine b-HCG (for all women between the age of 18 and 60 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperglycemia | up to 5 days of hospital course
  Defined as blood glucose > 180 mg/dL. This will be measured as the % of patient-days with a blood sugar > 180 mg/dL.

SECONDARY OUTCOMES:
Incidence of severe hyperglycemia | up to 5 days of hospital course
  Defined as blood glucose > 299 mg/dL. This will be measured as the % of patient-days with a blood sugar > 299 mg/dL.
Incidence of hypoglycemia | up to 5 days of hospital course
  Defined as blood glucose < 70 mg/dL. This will be measured as the % of patient-days with a blood sugar < 70 mg/dL.
Incidence of severe hypoglycemia | up to 5 days of hospital course
  Defined as blood glucose < 40 mg/dL. This will be measured as the % of patient-days with a blood sugar < 40 mg/dL.
Remission of primary oncologic diagnosis at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Garry Tobin, MD, Principal Investigator — Washington University School of Medicine; Anna Roshal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States